CLINICAL TRIAL: NCT06815536
Title: Master Protocol for Evaluating Multiple Infection Diagnostics for Ciprofloxacin-Resistant Neisseria Gonorrhoeae
Acronym: MASTERMINDRING
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); SpeeDx Pty Ltd (Industry); Abbott (Industry); Seegene USA Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00113379; UM1AI104681 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Neisseria Gonorrheae Infection
Keywords: mutant allele gyrA 91F; wildtype allele gyrA 91S; ciprofloxacin-resistant Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Urine: Investigational Reflex Test performed to detect the mutant gyrA 91F allele or the wildtype gyrA 91S allele using urine samples.
  Interventions: Diagnostic Test: Investigational Reflex Test 1; Diagnostic Test: Investigational Reflex Test 2; Diagnostic Test: Investigational Reflex Test 3
- Vaginal Swab: Investigational Reflex Test performed to detect the mutant gyrA 91F allele or the wildtype gyrA 91S allele using vaginal swabs.
  Interventions: Diagnostic Test: Investigational Reflex Test 1; Diagnostic Test: Investigational Reflex Test 2; Diagnostic Test: Investigational Reflex Test 3
- Pharyngeal Swabs: Investigational Reflex Test performed to detect the mutant gyrA 91F allele or the wildtype gyrA 91S allele using pharyngeal swabs.
  Interventions: Diagnostic Test: Investigational Reflex Test 1; Diagnostic Test: Investigational Reflex Test 2; Diagnostic Test: Investigational Reflex Test 3

INTERVENTIONS:
Diagnostic Test: Investigational Reflex Test 1 — Investigational Reflex Test 1
Diagnostic Test: Investigational Reflex Test 2 — Investigational Reflex Test 2
Diagnostic Test: Investigational Reflex Test 3 — Investigational Reflex Test 3

SUMMARY:
The goal of this study is to learn if a few investigational tests can correctly find the gene mutation (mutant allele gyrA 91F) that predicts ciprofloxacin resistance in clinical specimens that harbor Neisseria gonorrhoeae. The main question the study aims to answer:

Can the investigational reflex test find the correct gene mutation (Neisseria gonorrhoeae gyrA 91F or gyrA 91S) as compared to the sequenced result?

Specimens that are collected for routine clinical care and harbor Neisseria gonorrhoeae will be evaluated in this study.

DETAILED DESCRIPTION:
This is a prospective, multi-center, cross-sectional study using consecutive clinical specimens that are collected for routine clinical care and test positive for N. gonorrhoeae using an FDA-cleared molecular assay. The study evaluates the diagnostic accuracy of multiple investigational reflex tests to detect the mutant allele gyrA 91F that predicts ciprofloxacin resistance in N. gonorrhoeae, as compared to a reference standard of Sanger sequencing of the gyrA codon 91. Specimens will be tested via a reference standard of Sanger sequencing and one investigational reflex test. The target sample size is 311 urine specimens, 496 vaginal swab specimens, and 469 pharyngeal specimens, for each investigational reflex test.

ELIGIBILITY:
Inclusion Criteria:

* Be N. gonorrhoeae-positive on an FDA-cleared molecular assay
* Have sufficient N. gonorrhoeae-positive specimen volume for testing using the corresponding investigational reflex test and genetic sequencing
* Undergo proper handling and storage conditions

Exclusion Criteria:

* The N. gonorrhoeae-positive specimen media is not compatible with the investigational reflex test(s) at the laboratory site
* The N. gonorrhoeae-positive specimen is not clearly labeled by the laboratory to link to basic epidemiologic data (age, sex) and source

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical specimens from male and females that test positive for Neisseria gonorrhoeae
Sampling Method: Non-Probability Sample
Enrollment: 3291 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gyrA 91F identified by Investigational Reflex Test 1 relative to the sequenced results in urine | One day
  Investigational Reflex Test 1 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 1 relative to the sequenced results in vaginal swabs | One day
  Investigational Reflex Test 1 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 1 relative to the sequenced results in pharyngeal swabs | One day
  Investigational Reflex Test 1 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 2 relative to the sequenced results in urine | One day
  Investigational Reflex Test 2 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 2 relative to the sequenced results in vaginal swabs | One day
  Investigational Reflex Test 2 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 2 relative to the sequenced results in pharyngeal swabs | One day
  Investigational Reflex Test 2 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 3 relative to the sequenced results in urine | One day
  Investigational Reflex Test 3 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 3 relative to the sequenced results in vaginal swabs | One day
  Investigational Reflex Test 3 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.
Number of participants with gyrA 91F identified by Investigational Reflex Test 3 relative to the sequenced results in pharyngeal swabs | One day
  Investigational Reflex Test 3 results include gyrA 91F, gyrA 91S, invalid, and missing.
  Sanger Sequencing reference results include gyrA 91F, gyrA 91S, invalid, and missing.

SECONDARY OUTCOMES:
Number of invalid results for Investigational Reflex Test 1 in urine | One day
Number of invalid results for Investigational Reflex Test 1 in vaginal swabs | One day
Number of invalid results for Investigational Reflex Test 1 in pharyngeal swabs | One day
Number of invalid results for Investigational Reflex Test 2 in urine | One day
Number of invalid results for Investigational Reflex Test 2 in vaginal swabs | One day
Number of invalid results for Investigational Reflex Test 2 in pharyngeal swabs | One day
Number of invalid results for Investigational Reflex Test 3 in urine | One day
Number of invalid results for Investigational Reflex Test 3 in vaginal swabs | One day
Number of invalid results for Investigational Reflex Test 3 in pharyngeal swabs | One day

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Satlin, MD, MS, Principal Investigator — Weill Medical College of Cornell University; Jeffrey D. Klausner, MD, MPH, Principal Investigator — University of Southern California - Los Angeles; Vance G. Fowler, MD, MHS, Study Director — Duke University
Locations (8):
- United States (8):
  - San Francisco Public Health Laboratory, San Francisco, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Mississippi State Department of Public Health, Jackson, Mississippi
  - Corewell Health, Royal Oak, Missouri
  - LabCorp, Durham, North Carolina
  - ARUP Laboratories, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Molecular Testing Labs, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) including clinical specimen details, investigational testing results, and sequencing results can be shared with other researchers after primary publication. Investigators must apply to the Antibacterial Resistance Group for approval to receive and use the data. Investigators must comply with additional contractual and regulatory obligations.
Supporting Information: Study Protocol
Time Frame: IPD will be available after the primary publication date. There is not end date for the IPD availability.
Access Criteria: Only those who have applied to the ARLG and being approved will be able to access the data.
URL: https://arlg.org/request-data/